CLINICAL TRIAL: NCT01580930
Title: Changes in Physical Activity and Inactivity During a 12-week Exercise Training and/or Sedentary Time Intervention
Brief Title: Changes in Habitual Physical Activity and Inactivity
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kozey-Keadle; RC1HL099557 (NIH)
Record Dates: First submitted 2012-04-10; First posted 2012-04-19 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Habitual Physical Activity; Sedentary Time
Keywords: physical inactivity; exercise training; sedentary time; habitual physical activity
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group (No Intervention): Group had outcome measures collected and were instructed to not change activity and sedentary time behavior
- Exercise (Experimental): Participants performed 5 days per week, 40 min per session of exercise training under direct supervision of personal trainer.
  Interventions: Behavioral: exercise training
- Sedentary time reduction (Experimental): participants were give strategies to reduce sedentary time
  Interventions: Behavioral: sedentary time reduction
- exercise plus sedentary time reduction (Experimental): Participants completed exercise training (5 days per week, 40 min per session) plus were given sedentary time reduction intervention
  Interventions: Behavioral: exercsie training plus sedentary time reduction

INTERVENTIONS:
Behavioral: exercise training — 12 weeks, 5 days of week, 40 min per session of exercise training
  Arms: Exercise
Behavioral: sedentary time reduction — participants provided with strategies to decrease sitting
  Arms: Sedentary time reduction
Behavioral: exercsie training plus sedentary time reduction — 12 weeks of exercise training (5 days a week, 40 min per session) plus given strategies for reducing sitting time
  Arms: exercise plus sedentary time reduction

SUMMARY:
The purpose of this study is to determine if individuals involved in exercise training change habitual activity and inactivity behavior outside of exercise training. Eligible participants were randomly assigned to one of four groups: control, exercise training, sedentary time reduction, or exercise training plus sedentary time reduction. It was hypothesized that participants in the exercise training group will compensate for exercise training by reducing free-living physical activity behavior and increasing sedentary time. Participant free-living behavior was monitored for one week at baseline, 3, 6, 9 and 12 weeks using an activPAL wearable monitor.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants were those at increased risk of cardiovascular disease, based on meeting two of the following three criteria:

1. Pre-hypertensive: resting blood pressure between 125-160 mm Hg systolic and/or 85-100 mm Hg diastolic,
2. overweight/obese: body mass index (BMI) between 25 and 45 kg∙m-2,
3. high central adiposity: as defined by elevated natural waist circumference (> 102 cm [males] > 88cm [females]), a surrogate measure of visceral fat
4. low aerobic fitness (VO2 peak ≤ 50th percentile of age and sex specific norms)
5. exercising less than three days per week for less than 20 minutes per session for the preceding six months

Exclusion Criteria:

* major orthopedic limitations,
* wheelchair use or musculoskeletal problems that affected mobility,
* life-threatening illness (e.g., terminal cancer),
* chronic diseases (e.g., diagnosed heart disease, diabetes, emphysema) or
* any condition for which a physician did not recommend exercise. Participants were excluded if they had gastric bypass or lap-band surgery within the last year, were taking medication for type II diabetes (e.g. metformin) or beta-blocker medication for high blood pressure.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
change from baseline in sedentary time at 3 weeks | 3 weeks
  Measure is based on data collected with a wearable monitor that assesses time spent sitting/lying, standing, and walking
change from baseline in sedentary time at 6 weeks | 6 weeks
  Measure is based on data collected with a wearable monitor that assesses time spent sitting/lying, standing, and walking
change from baseline in sedentary time at 9 weeks | 9 weeks
  Measure is based on data collected with a wearable monitor that assesses time spent sitting/lying, standing, and walking
change from baseline in sedentary time at 12 weeks | 12 weeks
  Measure is based on data collected with a wearable monitor that assesses time spent sitting/lying, standing, and walking

SECONDARY OUTCOMES:
change from baseline in physical activity at 3 weeks | 3 weeks
  wearable monitor (activPAL) assesses number of steps, MVPA
change from baseline in physical activity at 6 weeks | 6 weeks
  wearable monitor (activPAL) assesses number of steps, MVPA
change from baseline in physical activity at 9 weeks | 9 weeks
  wearable monitor (activPAL) assesses number of steps, MVPA
change from baseline in physical activity at 12 weeks | 12 weeks
  wearable monitor (activPAL) assesses number of steps, MVPA

CONTACTS AND LOCATIONS:
Locations (1):
- UMass Amherst Physical Activity and Health Lab, Amherst, Massachusetts, United States